CLINICAL TRIAL: NCT02043301
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, PARALLEL GROUP STUDY TO ASSESS INJECTION SITE RELATIVE BIOAVAILABILITY OF PF-04950615 FOLLOWING SUBCUTANEOUS ADMINISTRATION IN ADULT SUBJECTS WITH HYPERCHOLESTEROLEMIA
Brief Title: Pharmacokinetics And Relative Bioavailability Of Bococizumab (PF-04950615; RN316) When Administered To The Abdomen, Thigh Or Upper Arm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1481024
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Hypercholesterolemia
Keywords: pharmacokinetics; bioavailability; PF-04950615
MeSH Terms: conditions — Hypercholesterolemia | interventions — bococizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single 150 mg PF-04950615 dose administered to the abdomen (Active Comparator)
  Interventions: Biological: Bococizumab (PF-04950615; RN316)
- Single 150 mg PF-04950615 dose administered to the upper arm (Experimental)
  Interventions: Biological: Bococizumab (PF-04950615; RN316)
- Single 150 mg PF-04950615 dose administered to the thigh (Experimental)
  Interventions: Biological: Bococizumab (PF-04950615; RN316)

INTERVENTIONS:
Biological: Bococizumab (PF-04950615; RN316) — Single 150 mg PF-04950615 dose administered SC to the abdomen
  Arms: Single 150 mg PF-04950615 dose administered to the abdomen
Biological: Bococizumab (PF-04950615; RN316) — Single 150 mg PF-04950615 dose administered SC to the upper arm
  Arms: Single 150 mg PF-04950615 dose administered to the upper arm
Biological: Bococizumab (PF-04950615; RN316) — Single 150 mg PF-04950615 dose administered SC to the thigh
  Arms: Single 150 mg PF-04950615 dose administered to the thigh

SUMMARY:
This study aims to characterize the single dose pharmacokinetics of PF-04950616 following subcutaneous injection to the abdomen, upper arm or the thigh.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age.
* Body Mass Index (BMI) ≤ 33 kg/m2, and total body weight of 60 kg to 90 kg (132 lbs to 198 lbs).
* Fasting LDL-C must be > 130 mg/dL (borderline high per NCEP ATP III criteria) at two qualifying visits: initial screening (Days -28 to -14) and Day -7.

Exclusion Criteria:

* Poorly controlled type 1 or type 2 diabetes mellitus (HbA1c > 9.0%).
* History of a cardiovascular or cerebrovascular event (eg, MI, stroke, TIA) or related procedure (eg, angioplasty) during the past year.
* Subjects who meet the New York Heart Association (NYHA) criteria for congestive heart failure (CHF) classes III or IV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Wang EQ, Plotka A, Salageanu J, Sattler C, Yunis C. Pharmacokinetics and pharmacodynamics of bococizumab, a monoclonal antibody to PCSK9, after single subcutaneous injection at three sites [NCT 02043301]. Cardiovasc Ther. 2017 Oct;35(5). doi: 10.1111/1755-5922.12278. PMID 28636184
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481024&StudyName=Pharmacokinetics%20And%20Relative%20Bioavailability%20Of%20PF-04950615%20When%20Administered%20To%20The%20Abdomen%2C%20Thigh%20Or%20Upper%20Arm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy-five (75) participants were enrolled and randomized in a 1:1:1 ratio to receive a single dose of Treatment A (PF-04950615 [hereafter referred to as bococizumab] 150 mg subcutaneously [SC] to the abdomen), Treatment B (bococizumab 150 mg SC to the thigh), or Treatment C (bococizumab 150 mg SC to the upper arm).
Groups:
- Bococizumab 150 mg Abdomen: Participants received a single dose of bococizumab 150 mg SC to the abdomen.
- Bococizumab 150 mg Thigh: Participants received a single dose of bococizumab 150 mg SC to the thigh.
- Bococizumab 150 mg Upper Arm: Participants received a single dose of bococizumab 150 mg SC to the upper arm.
Period: Overall Study
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Started | 25 | 25 | 25
Completed | 25 | 24 | 25
Not Completed | 0 | 1 | 0
Not completed — Discontinued | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 0 (11.7) | 0 (7.5) | 0 (9.6) | 0
  18-44 years | 11 | 7 | 8 | 26
  45-64 years | 13 | 18 | 17 | 48
  Greater than or equal to (>=) 65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 13 | 35
  Male | 15 | 13 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: AUCinf is the area under the plasma concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time.
Time Frame: Day 1 (Hour 0 pre-dose, Hours 1 and 8 post-dose), Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, Day 57, Day 64, Day 71 and Day 85/Early Termination.
Population: The pharmacokinetic (PK) parameter analysis population included all enrolled participants who received at least 1 dose of study medication and that had at least 1 of the PK parameters of interest. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (mcg*day/mL)
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 24 | 25 | 25
micrograms*day/milliliter (mcg*day/mL) | 175.9 (53) | 198.9 (30) | 160.3 (33)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Thigh (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 120.96, 90% CI 2-sided [101.99 to 143.45]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Upper Arm (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 94.93, 90% CI 2-sided [80.20 to 112.38]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed concentration.
Time Frame: as for outcome 1
Population: The PK parameter analysis population included all enrolled participants who received at least 1 dose of study medication and that had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
mcg/mL | 9.68 (51) | 11.89 (30) | 8.14 (32)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Thigh (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 127.65, 90% CI 2-sided [107.19 to 152.02]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Upper Arm (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 86.16, 90% CI 2-sided [72.49 to 102.40]

3. Secondary Outcome: Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast)
Description: AUClast is area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
mcg*day/mL | 158.8 (65) | 192.5 (31) | 152.6 (36)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Thigh (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 129.98, 90% CI 2-sided [106.76 to 158.27]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Upper Arm (Test) versus Abdomen (Reference); Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed body weight as a covariate; Adjusted Geometric Means Ratio (%) = 100.27, 90% CI 2-sided [82.54 to 121.82]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Time for maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
days | 5.04 [2.00 to 7.02] | 4.25 [2.92 to 6.97] | 6.93 [2.00 to 14.1]

5. Secondary Outcome: Apparent Clearance (CL/F)
Description: Apparent clearance following subcutaneous administration.
Time Frame: as for outcome 1
Population: The PK parameter analysis population included all enrolled participants who received at least 1 dose of study medication and that had at least 1 of the PK parameters of interest. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per day
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 24 | 25 | 25
liters per day | 0.8521 (53) | 0.7545 (30) | 0.9352 (33)

6. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Apparent volume of distribution following subcutaneous administration.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 24 | 25 | 25
liters | 8.84 (49) | 7.98 (29) | 11.33 (36)

7. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: Terminal elimination half-life following subcutaneous administration.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 24 | 25 | 25
days | 7.27 (1.09) | 7.40 (1.03) | 8.53 (1.61)

8. Secondary Outcome: Maximum Low-density Lipoprotein Cholesterol LDL-C Lowering Effect (Emax): Absolute Value
Description: Maximum LDL-C response using absolute on trial LDL-C data
Time Frame: Baseline (average of Day -7 and Day 1), Day 2, Day 3, Day 4, Day 5, Day 6, Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, Day 57, Day 64, Day 71 and Day 85/Early Termination
Population: The pharmacodynamic (PD) analysis population included all enrolled participants who received at least 1 dose of study medication and had both baseline and post-baseline values for at least 1 of the PD endpoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
mg/dL | 72.20 (20.185) | 75.32 (31.964) | 74.40 (25.290)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 97.35, 90% CI 2-sided [84.659 to 111.943]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 103.96, 90% CI 2-sided [90.405 to 119.557]

9. Secondary Outcome: Emax: Change From Baseline
Description: LDL-C Emax expressed as change from baseline.
Time Frame: as for outcome 8
Population: The PD analysis population included all enrolled participants who received at least 1 dose of study medication and had both baseline and post-baseline values for at least 1 of the PD endpoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
mg/dL | -96.88 (19.356) | -97.62 (26.967) | -90.46 (25.441)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 97.10, 90% CI 2-sided [86.558 to 108.926]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 93.52, 90% CI 2-sided [83.359 to 104.912]

10. Secondary Outcome: Emax: Percent Change From Baseline
Description: LDL-C Emax expressed as percent change from baseline.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
percent change | -57.47 (9.084) | -56.98 (14.740) | -54.96 (13.269)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 97.10, 90% CI 2-sided [86.558 to 108.926]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 93.52, 90% CI 2-sided [83.359 to 104.912]

11. Secondary Outcome: Time to Reach Maximum LDL-C Lowering (Tmax, LDL-C)
Description: Time to LDL-C Emax
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
days | 20.96 (7.461) [5.0 to 34.1] | 20.06 (5.173) [4.2 to 28.0] | 14.01 (7.102) [7.1 to 42.0]

12. Secondary Outcome: Area Under the LDL-C Effect Curve (AUEC): Absolute Value
Description: AUEC is the area under the LDL-C concentration-time curve from baseline to Day 85 exprssed using absolute on trial value
Time Frame: as for outcome 8
Population: The PD analysis population included all enrolled participants who received at least 1 dose of study medication and had both baseline and post-baseline values for at least 1 of the PD endpoints. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mg*day/dL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 24 | 25
mg*day/dL | 11181.64 (1545.335) | 11682.39 (2063.772) | 11231.39 (1928.904)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 102.51, 90% CI 2-sided [97.555 to 107.717]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 102.02, 90% CI 2-sided [97.131 to 107.151]

13. Secondary Outcome: AUEC: Change From Baseline
Description: AUEC is the area under the LDL-C concentration-time curve from baseline to Day 85 exprssed as change from baseline
Time Frame: as for outcome 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg*day/dL
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 24 | 25
mg*day/dL | -2982.16 (1431.589) | -2701.99 (1432.539) | -2546.68 (977.934)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 79.09, 90% CI 2-sided [60.883 to 102.735]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 91.15, 90% CI 2-sided [70.269 to 118.248]

14. Secondary Outcome: AUEC: Percent Change From Baseline
Description: AUEC is the area under the LDL-C concentration-time curve from baseline to Day 85 expressed as percent change from baseline.
Time Frame: as for outcome 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 24 | 25
percent change | -1715.22 (758.720) | -1538.85 (724.925) | -1550.73 (583.745)
Statistical Analysis 1: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Thigh; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 79.09, 90% CI 2-sided [60.883 to 102.735]
Statistical Analysis 2: Comparison: Bococizumab 150 mg Abdomen vs Bococizumab 150 mg Upper Arm; Test type: Superiority or Other — Ratios (and 90% confidence intervals) were expressed as percentages; ANCOVA; ANCOVA model with treatment group as a fixed effect and log-transformed baseline LDL-C as a covariate; Adjusted Geometric Means Ratio (%) = 91.15, 90% CI 2-sided [70.269 to 118.248]

15. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) by Severity
Description: Acute injection site reactions (e.g, pain, pruritus, induration) were captured as adverse events (AEs). Intensity of the AE was described as mild (does not interfere with usual function), moderate (interferes to some extent with usual function), or severe (interferes significantly with participant's usual function).
Time Frame: Day 1 to Day 85
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
participants
  Mild: injection site erythema | 1 | 0 | 2
  Mild: injection site indurations | 1 | 2 | 0
  Mild: injection site pain | 1 | 0 | 0
  Mild: injection site pruritus | 0 | 0 | 1
  Mild: injection site reaction | 1 | 3 | 1
  Mild: injection site swelling | 0 | 1 | 0
  Moderate: injection site erythema | 0 | 0 | 0
  Moderate: injection site indurations | 0 | 0 | 0
  Moderate: injection site pain | 0 | 0 | 0
  Moderate: injection site pruritus | 0 | 0 | 0
  Moderate: injection site reaction | 0 | 0 | 0
  Moderate: injection site swelling | 0 | 0 | 0
  Severe: injection site erythema | 0 | 0 | 0
  Severe: injection site indurations | 0 | 0 | 0
  Severe: injection site pain | 0 | 0 | 0
  Severe: injection site pruritus | 0 | 0 | 0
  Severe: injection site reaction | 0 | 0 | 0
  Severe: injection site swelling | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb)
Description: A participant is ADA positive if ADA titer (log2) >=6.23. A participant is nAb positive if nAb titer (log2) >=4.32.
Time Frame: Day 1, Day 15, Day 29, Day 57 and Day 85/Early Termination
Population: The safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
participants
  Positive ADA | 6 | 6 | 11
  Positive nAb | 2 | 2 | 0

17. Secondary Outcome: Anti-Drug Antibody (ADA) Titer
Description: ADA titer: titers were presented as log2 reciprocal dilution at assay cutpoint.
Time Frame: Day 1, Day 15, Day 29, Day 57 and Day 85/Early Termination
Population: The safety analysis population included all participants who received at least 1 dose of study medication. Only confirmed ADA positive samples were analyzed for titer.
Measure: Median (Full Range); unit: Log2 titer
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Number analyzed (Participants) | 25 | 25 | 25
Log2 titer
  Day 15: number analyzed (Participants) | 1 | 1 | 0
  Day 15 | NA [13.65 to 13.65] — Only 1 participant has reportable data, median value is not applicable. | NA [7.91 to 7.91] — Only 1 participant has reportable data, median value is not applicable. |
  Day 29: number analyzed (Participants) | 1 | 2 | 0
  Day 29 | NA [12.49 to 12.49] — Only 1 participant has reportable data, median value is not applicable. | NA [6.23 to 7.39] — Only 2 participants have reportable data, median value is not applicable. |
  Day 57: number analyzed (Participants) | 1 | 3 | 4
  Day 57 | NA [13.22 to 13.22] — Only 1 participant has reportable data, median value is not applicable. | 7.64 [7.61 to 10.84] | 8.25 [6.35 to 9.28]
  Day 85: number analyzed (Participants) | 6 | 5 | 11
  Day 85 | 7.46 [6.31 to 13.57] | 7.20 [6.23 to 15.05] | 7.60 [6.23 to 13.01]

18. Secondary Outcome: Neutralizing Antibody (nAb) Titer
Description: nAb titer: titers were presented as log2 reciprocal dilution at assay cutpoint.
Time Frame: Day 1, Day 15, Day 29, Day 57 and Day 85/Early Termination
Population: The safety analysis population included all participants who received at least 1 dose of study medication. Only confirmed ADA positive samples were analyzed for nAb. nAb titer was determined if a sample is screened positive for nAb. nAb titer data for the Bococizumab 150 mg Upper Arm group is not presented as there were no nAb positive subjects.
Measure: Median (Full Range); unit: Log2 titer
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh
Number analyzed (Participants) | 25 | 25
Log2 titer
  Day 29: number analyzed (Participants) | 1 | 0
  Day 29 | NA [6.24 to 6.24] — Only 1 participant has reportable data, median value is not applicable. |
  Day 57: number analyzed (Participants) | 1 | 1
  Day 57 | NA [5.93 to 5.93] — Only 1 participant has reportable data, median value is not applicable. | NA [4.94 to 4.94] — Only 1 participant has reportable data, median value is not applicable.
  Day 85: number analyzed (Participants) | 2 | 2
  Day 85 | NA [4.40 to 6.03] — Only 2 participants have reportable data, median value is not applicable. | NA [4.32 to 7.35] — Only 2 participants have reportable data, median value is not applicable.

ADVERSE EVENTS:
Time Frame: Baseline up to Day 85
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Bococizumab 150 mg Abdomen | Bococizumab 150 mg Thigh | Bococizumab 150 mg Upper Arm
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 13/25 | 15/25 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bococizumab 150 mg Abdomen (N=25) | Bococizumab 150 mg Thigh (N=25) | Bococizumab 150 mg Upper Arm (N=25)
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bococizumab 150 mg Abdomen (N=25) | Bococizumab 150 mg Thigh (N=25) | Bococizumab 150 mg Upper Arm (N=25)
Noninfective conjunctivitis (Eye disorders) | 0 | 0 | 1
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 1 | 0 | 2
Injection site induration (General disorders) | 1 | 2 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 3 | 1
Injection site swelling (General disorders) | 0 | 1 | 0
Therapeutic response changed (General disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.